CLINICAL TRIAL: NCT03622801
Title: Risk of Anaphylactoid Reactions of Iopromide After Intra-arterial Administration
Brief Title: Study on the Risk of Allergy-like Reactions After Intra-arterial or Intra-venous Injection of the Marketed X-ray Contrast Medium Iopromid
Acronym: UVIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19677
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Contrast Medium
MeSH Terms: interventions — iopromide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intra-arterial administration: Patients with intra-arterial administration of Iopromide
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)
- Intravenous administration: Patients with intravenous administration of Iopromide
  Interventions: Drug: Iopromide (Ultravist, BAY86-4877)

INTERVENTIONS:
Drug: Iopromide (Ultravist, BAY86-4877) — Patients who have received Iopromide (iodine concentrations of 300 mg/mL or 370 mg/mL) either intra-venously or intra-arterially.

SUMMARY:
Iopromide (trade name is Ultravist) is on the market for more than 30 years and has been used more than 250 million times as X-ray contrast medium for patients. It is known that Iopromide may cause allergy-like reactions after being injected. With this study researchers want to find out, if the risk of severe allergy-like reactions is lower, when Iopromide will be injected into an artery, compared to the risk after an injection of Iopromid into a vein. To find this out data from four trials on Iopromide that are already completed will be combined and newly analyzed. The database used for this analysis will contain data from more than 150,000 patients.

ELIGIBILITY:
The study population consists of patients who received a contrast enhanced x-ray examination with Iopromide for various clinical reasons. Iopromide was administered either intra-venously or intra-arterially.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who received a contrast enhanced x-ray examination with Iopromide for various clinical reasons. Iopromide was administered either intra-venously or intra-arterially.
Sampling Method: Non-Probability Sample
Enrollment: 133331 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with anaphylactoid reactions of Iopromide after administration | Retrospective analysis from 31 Aug 2010 to 30 Sep 2011

SECONDARY OUTCOMES:
Number of patients with anaphylactoid reactions after intra-arterial administration of Iopromide | Retrospective analysis from 31 Aug 2010 to 30 Sep 2011
Number of patients with anaphylactoid reactions after intra-venous administration of Iopromide | Retrospective analysis from 31 Aug 2010 to 30 Sep 2011

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Germany